CLINICAL TRIAL: NCT01349543
Title: The Development of a Human Model of Respiratory Syncytial Virus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JROSM0127
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Syncytial Virus Infections; Respiratory Viral Infections
Keywords: Respiratory syncytial virus; RSV; Immunology; Viral infection; Bronchiolitis; Viral challenge; Viral lung disease
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases; Bronchiolitis | interventions — beta-lactamase CTX-M-37, Salmonella enterica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Viral Challenge (Experimental)
  Interventions: Biological: RSV A Memphis 37

INTERVENTIONS:
Biological: RSV A Memphis 37 — Intranasal administration
  Other Names: M37

SUMMARY:
The aim of this study is to understand the immune response (how the body fights infection) to Respiratory Syncytial Virus (RSV). This virus usually causes a simple 'common cold' illness in healthy adults, but can cause wheezing and lung problems in young infants and the elderly. The investigators want to understand why this is, in order to develop vaccines and treatments.

Participants will include 30-40 healthy adults age 18-55 years. Study procedures will include brief medical exams, breathing tests, a diary of symptoms, blood tests, samples of fluid (lavage) and cells from the nose, throat and lungs. All participants will receive the virus via drops in the nose. The duration of the study for all subjects will be 6 weeks.

DETAILED DESCRIPTION:
Bronchiolitis is the commonest cause of hospital admission in infants. It is caused by Respiratory Syncytial Virus(RSV), a virus that causes mild 'common colds' in adults, but can cause lung inflammation and difficulty breathing in infants and the elderly. In 2005, nearly 34 million cases in children <5 years occurred, resulting in 3.4 million hospital admissions,and around 120,000 deaths. There is no vaccine, and some previous vaccines actually made the disease worse.

The investigators have been trying to understand why for 40 years. Advances in immunology have given us a completely different way of looking at inflammation: rather than studying what causes it, the investigators now want to know what regulates it. Much of what the investigators know about how what causes and regulates inflammation has come from studies of animals, however, these do not exactly predict what happens in man.

The investigators therefore plan to infect healthy adult volunteers with RSV, and observe what happens in humans after RSV infection. The investigators will collect samples of blood, fluid and cells from the nose, throat, and lungs, and a diary of symptoms over four weeks. The investigators will analyse the blood, fluid, and cells to determine the important mechanisms that regulate inflammation in human RSV infection.

Studies like this have been conducted previously with no severe side effects. The investigators anticipate that the discoveries made in this research project will help us achieve a better understanding of what causes and regulates inflammation in RSV so that the investigators can learn ways to control it, with the aim of developing vaccines and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 18 to 55 years, able to give informed consent

Exclusion Criteria:

* Chronic respiratory disease (asthma, COPD, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 6 months
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Smoking in the past 6 months OR >5 pack-year lifetime history
* Subjects with allergic symptoms present at baseline
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Subjects with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by the study doctor to make the participant unsuitable for the study
* Pregnant or breastfeeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Openshaw, Principal Investigator — Imperial College London
Locations (1):
- St. Mary's Hospital, Imperial College London, Norfolk Place,, London, United Kingdom

REFERENCES:
- [Result] Habibi MS, Thwaites RS, Chang M, Jozwik A, Paras A, Kirsebom F, Varese A, Owen A, Cuthbertson L, James P, Tunstall T, Nickle D, Hansel TT, Moffatt MF, Johansson C, Chiu C, Openshaw PJM. Neutrophilic inflammation in the respiratory mucosa predisposes to RSV infection. Science. 2020 Oct 9;370(6513):eaba9301. doi: 10.1126/science.aba9301. PMID 33033192

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Viral Challenge
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Viral Challenge
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not used as a baseline measure.
  Participants
    Female | 21
    Male | 37
Region of Enrollment [Number; unit: participants]
  United Kingdom | 58
Assessed as healthy with no pre-existing disease [Count of Participants; unit: Participants] | 58

OUTCOME MEASURES:

1. Primary Outcome: Host Response to RSV Challenge Measured as Change From Baseline of Chemical Mediators in Nasal Fluid
Description: The host response to RSV challenge has been assessed at baseline, daily for 14 days and at study conclusion (28 days) using methods such as symptom diaries, volume of nasal secretions, numbers of inflammatory cells in nasal mucus, and levels of chemical mediators in nasal fluids.
Time Frame: Prior to and 0-28 days post challenge
Measure: Count of Participants; unit: Participants
Groups:
- Viral Challenge; Resulting in Common Cold Symptoms: RSV A Memphis 37: Intranasal administration resulting in a cold
Arm/Group | Viral Challenge; Resulting in Common Cold Symptoms
Number analyzed (Participants) | 58
Participants | 23

ADVERSE EVENTS:
Groups:
- Viral Challenge; Common Cold Symptoms: RSV A Memphis 37: Intranasal administration resulting in common cold
Arm/Group | Viral Challenge; Common Cold Symptoms
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes